CLINICAL TRIAL: NCT01718379
Title: A Phase II Study Evaluating the Efficacy/Safety of Lenalidomide With or Without Epoetin Beta in Transfusion-dependent ESA-resistant Patients With IPSS Low- and Intermediate-1 Risk Myelodysplastic Syndromes Without Chromosome 5 Abnormality.
Brief Title: Lenalidomide in Subject With Low and Intermediate-1 Risk MDS and Without Chromosome 5 Abnormality.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Celgene (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM-Len-Epo-08
Record Dates: First submitted 2012-10-23; First posted 2012-10-31 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplasia
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — Lenalidomide; epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Lenalidomide 10 mg/day for 21 days every 28 days for 4 courses.
  Evaluation of response at the end of 4 months according to IWG 2006 and IWG 2000 criteria.
  Maintenance: responders will continue to follow the corresponding treatment arm until relapse occurs; non responders at cycle 4 in arm A will be considered in failure of treatment and the introduction of Epoetin beta is at the discretion of the physician.
  The patients will be followed every 3 months for 12 months
  Interventions: Drug: Lenalidomide
- Arm B (Experimental): Lenalidomide 10 mg/day for 21 days every 28 days for 4 courses combined with weekly subcutaneous injections of Epoetin beta (60,000 Units/w).
  Evaluation of response at the end of 4 months according to IWG 2006 and IWG 2000 criteria.
  Maintenance: responders will continue to follow the corresponding treatment arm until relapse occurs; non responders at cycle 4 in arm A will be considered in failure of treatment and the introduction of Epoetin beta is at the discretion of the physician.
  The patients will be followed every 3 months for 12 months
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide:10 mg per day during 21 days
  Other Names: Revlimid
  Arms: Arm A
Drug: Epoetin beta — Epoetin beta: 60,000 Units/week.
  Other Names: NEORECORMON
  Arms: Arm B

SUMMARY:
The goal of the present study is to assess, through a randomized phase II trial, the efficacy and safety of Lenalidomide with or without Epoetin beta in transfusion-dependent, ESA-resistant, IPSS low and intermediate-1 risk MDS patients without chromosome 5 abnormality.

Patients will receive either Lenalidomide alone or Lenalidomide and Epoetin beta for 4 months. Responders will be eligible for maintenance treatment with cycles identical to the first cycles, until relapse occurs or until unacceptable toxicity.

DETAILED DESCRIPTION:
This is a multi-center, open-label, randomized, Phase II study.

Patients will be treated either with arm A or B

* Arm A: Lenalidomide 10 mg/day for 21 days every 28 days for 4 courses.
* Arm B: Lenalidomide 10 mg/day for 21 days every 28 days for 4 courses combined with weekly subcutaneous injections of Epoetin beta (60,000 Units/w).

Evaluation of response at the end of 4 months according to IWG 2006 and IWG 2000 criteria.

Maintenance: responders will continue to follow the corresponding treatment arm until relapse occurs; non responders at Evaluation of response at the end of 4 months according to IWG 2006 and IWG 2000 criteria.

in arm A will be considered in failure of treatment and the introduction of Epoetin beta is at the discretion of the physician.

The patients will be followed every 3 months for 12 months

ELIGIBILITY:
Inclusion Criteria:

MDS defined as

* Low or int-1 IPSS score
* Documented absence of chromosome 5 abnormality (del(5q) or -5 karyotype)
* De novo MDS, excluding therapy-related MDS AND
* Transfusion dependance (requirement of at least 4 units of RBC transfusions every 8 weeks )
* Resistance or loss of response to a previous treatment with Epoetin alpha/beta (at least 60,000 Units/w) or Darbepoetin (at least 250 µg/w), for at least 12 weeks
* Ineligibility for allogeneic stem cell transplantation or intensive chemotherapy during the next 12 months
* ECOG performance status ≤ 2
* Age ≥ 18 years
* Life expectancy ≥ 3 months
* Adequate liver function (transaminases serum levels ≤ 3N)
* Adequate renal function (calculate creatinine clearance > 50 ml/min)
* Female subjects of chilbearing potential* must :

Agree to use effective contraception without interruption throughout the study and for at least 4 weeks after the end of treatment

• Men must: Agree to not conceive during the treatment and to use effective contraception during the treatment period (including periods of dose reduction or temporary suspension) and during one week after end of treatment if their partner is of childbearing potential.

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics
* Platelets less than 50 G/L
* Prior history of deep vein thrombosis or pulmonary embolism
* Previous treatment by Thalidomide
* Treatment with any investigational antileukemic agent or chemotherapy at least 6 weeks prior to study entry and lack of full recovery from side effects due to prior therapy independent of when that therapy were given
* Rapidely progressive disease with copromised organ function judged to be life-threatening by the Investigator
* Pregnant or lactating female
* Known human immunodeficiency virus (HIV) infection
* Known active hepatitis B and/or C virus infection
* Hypersensitivity or intolerance to Lenalidomide or any of the excipients
* Hypersensitivity to Epoetin beta or any of the excipients
* Uncontrolled arterial hypertension
* Any history of malignancy (other than myelodysplastic syndrome) unless the patient has remained disease free for more than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Comparing the efficacy of Lenalidomide alone to Lenalidomide with Epoetin beta in transfusion-dependent ESA-resistant | After 4 months of treatment
  Primary outcome is a complete or partial response defined by the IWG 2006 criteria observed after 4 months of treatment. Comparison in the rate of response between the two groups will be performed with Chi-square test or if necessary Fisher exact test.
  Same analyzes will be performed with the IWG 2000 response definition .

SECONDARY OUTCOMES:
will be to assess the safety of Lenalidomide and of its combination with Epoetin beta | After 2 months of treatment
  * Safety of Lenalidomide and of its combination with Epoetin beta: adverse events (type, frequency, severity) and relationship of adverse events to study drug
  * % of major HI-E and minor HI-E after 4 courses according to IWG 2000 criteria
  * Erythroid response duration
  * Time to response
  * Time to progression according to IPSS
  * RBC transfusion independence
  * Prognostic factors of response
  * Survival
  * Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Andréa TOMA, MD, Principal Investigator — Groupe Francophone des Myelodysplasies; François Dreyfus, MD, Study Director — Groupe Francophone des Myelodysplasies
Locations (48):
- France (47):
  - Hematology Dpt, Service d'Hématologie Clinique, CHU Albert Michallon, Grenoble
  - Hematology Dpt, CHR La Source orléans, Orléans, Orléans
  - Chu Amiens, Amiens
  - CHU Angers, Angers
  - Hematology Dpt, CH d'Avignon-305 rue Follereau-, Avignon
  - CH de la Cote Basque, Bayonne
  - centre de Blois, Blois
  - Hopital Avicenne, Bobigny
  - Hematology Dpt, CHU Haut-Lévèque, Bordeaux
  - Hôpital Boulogne Sur Mer, Boulogne-sur-Mer
  - hôpital Morvan, Brest
  - CHU Clémenceau, Caen
  - CH de Carcassonne, Carcassonne
  - Hematology Dpt, CH René Dubos, Cergy-Pontoise
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH de Compiègne, Compiègne
  - Hematology Dpt, Hôpital Sud Francilien, Corbeil-Essonnes
  - hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - Hematology Dpt, Hôpital Versailles, Le Chesnay
  - Hematology Dpt,CH Le mans, Le Mans
  - CHRU Huriez, Lille
  - Hopital Saint-Vincent de Paul, Lille
  - CHRU de Limoges, Limoges
  - Hematology Dpt, Centre Hospitalier Lyon Sud, Lyon
  - CH de Mantes-la-jolie, Mantes-la-Jolie
  - Institut Paoli Calmettes, Marseille
  - Hematology Dpt, CHU Brabois, Nancy
  - Hematology Dpt, CHU de nantes, Nantes
  - Hematology Dpt, CHU Archet, Nice
  - Hematology Dpt, CHU Caremeau, Nîmes
  - Hematology Dpt, Hôpital la pitié-Salpétrière, Paris
  - Hematology Dpt, Hopital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - centre René Huguenin, Paris Saint Cloud
  - Hematology Dpt, Hôpital Maréchal Joffre, Perpignan
  - Hôpital Jean Bernard, Poitiers
  - Hematology Dpt, Centre Hospitalier de la région d'Annecy, Pringy
  - CHRU de Reims, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CH de Saint Quentin, Sint Quentin
  - Chu Strasbourg, Strasbourg
  - Hematology Dpt, CHU PURPAN, Toulouse
  - Hematology Dpt, CH CHU Bretoneau, Tours
  - Hematology Dpt, CHU de Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
  - Hematology Dpt, CHU Cochin, Paris, Île-de-France Region
- centre hopitalier princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chesnais V, Renneville A, Toma A, Lambert J, Passet M, Dumont F, Chevret S, Lejeune J, Raimbault A, Stamatoullas A, Rose C, Beyne-Rauzy O, Delaunay J, Solary E, Fenaux P, Dreyfus F, Preudhomme C, Kosmider O, Fontenay M; Groupe Francophone des Myelodysplasies. Effect of lenalidomide treatment on clonal architecture of myelodysplastic syndromes without 5q deletion. Blood. 2016 Feb 11;127(6):749-60. doi: 10.1182/blood-2015-04-640128. Epub 2015 Dec 1. PMID 26626993